CLINICAL TRIAL: NCT05767138
Title: Knowledge, Attitudes, Practices and Willingness to Vaccinate in Preparation for the Introduction of HPV Vaccines in Bamako, Mali
Brief Title: STI Knowledge and HPV Vaccine Acceptance in Bamako, Mali in 2012
Status: Completed | Type: Observational
Sponsor: Global Alliance to Immunize Against AIDS Vaccine Foundation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HPV Vaccine Survey
Record Dates: First submitted 2022-10-26; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: HPV; HPV-Related Cervical Carcinoma
Keywords: Mali; Bamako; Survey

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bamako Participants: 301 male and female participants. Teenagers and adults. Living in two urban regions of Bamako.
  Interventions: Behavioral: HPV Vaccine Acceptance Survey

INTERVENTIONS:
Behavioral: HPV Vaccine Acceptance Survey

SUMMARY:
Although screening for pre-cancerous cervical lesions and human papilloma virus (HPV) vaccination are accepted and effective means to prevent cervical cancer, women in Mali have limited access to these interventions. In addition, cervical cancer prevention by HPV vaccination has been controversial in some settings. To reduce cervical cancer prevalence and increase HPV vaccine uptake, it is important to understand the level of knowledge about cervical cancer screening and practices related to vaccination in at-risk populations. In this study, the level of knowledge about HPV and cervical cancer and attitudes towards vaccination were assessed among 301 participants (male and female, adults and adolescents) in a house-to-house survey in two urban neighborhoods in Bamako, Mali. The survey was combined with a brief educational session on HPV. Prior to the education session, overall knowledge of HPV infection and cervical cancer was very low: only 8% knew that HPV is a sexually transmitted infection (STI). Less than 20% of women had ever consulted a gynecologist and less than 3% had ever had cervical cancer screening. After hearing a description of HPV vaccine, more than 80% would accept HPV vaccination; fathers and husbands were identified as primary decisions makers and local clinics or the home as preferred sites for vaccination. This study provides information on STI knowledge and vaccine acceptance in Bamako, Mali in 2012, prior to the introduction of HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years of age, with guardian consent
* 18 years or older
* Male or Female
* Living in Mèkin-Sikoro and Djikoroni

Exclusion Criteria:

* 12-17 years of age, without guardian consent
* <12 years of age
* Living outside Mèkin-Sikoro and Djikoroni

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants were recruited between May and June 2011 in Mèkin-Sikoro and Djikoroni, two peri-urban communities of Bamako that have been site for previous population surveys. Adolescents were eligible if aged 12-17 years and living in the household, and if a guardian was available to provide consent. Adults (male and female) were eligible if aged >18 years and living in the household. A total of 301 participants participated (150 living in households in Djikoroni, 151 living in Me´kin-Sikoro)
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Participants' acceptance of the vaccine | immediately after the intervention
  Number of participants willing to be vaccinated against HPV and their vaccination preferences after educational sessions

SECONDARY OUTCOMES:
Knowledge of STIs, HPV, and Cervical Cancer | immediately after the intervention
  Knowledge Question asked before and after educational session

CONTACTS AND LOCATIONS:
Overall Officials: Anne De Groot, MD, Principal Investigator — GAIA Vaccine Foundation

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-03-18): https://cdn.clinicaltrials.gov/large-docs/38/NCT05767138/Prot_SAP_ICF_000.pdf